CLINICAL TRIAL: NCT00267124
Title: KU Brain Aging Project
Brief Title: Brain Aging Project--Kansas University
Status: Completed | Type: Observational
Sponsor: University of Kansas Medical Center (Other)
Collaborators: University of Kansas (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Other Study IDs: IA0089; 1R03AG026374-01 (NIH)
Record Dates: First submitted 2005-12-16; First posted 2005-12-20 (Estimated); Last update posted 2017-04-06 (Actual); Status verified 2017-04

CONDITIONS: Alzheimer's Disease
Keywords: cognitive decline; dementia; neuroimaging
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction; Dementia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples are collected analyzed and banked as whole blood, serum, white blood cells

GROUPS / COHORTS (2):
- 1: elderly people who have normal cognition
- 2: elderly people who have mild to moderate Alzheimer's disease

SUMMARY:
The purpose of this study is to determine the effects of exercise and cardiorespiratory fitness on age-related brain changes.

DETAILED DESCRIPTION:
The mission of the KU Brain Aging Project is to promote healthy brain aging. How the brain changes with age is not well-characterized and even less is known about the factors influencing the rate of brain aging. Thus, we are using MRI scans to examine the structure of the brain in relation to important lifestyle factors. This will allow us to better understand the processes influencing the brain as it ages. In turn, this will help identify specific ways to promote healthy brain aging and, perhaps, prevent the onset of Alzheimer's disease.

Participants complete 4 visits over several months. The first visit entails a clinical evaluation and memory testing involving the use of paper and pencil testing. The second visit is an MRI brain scan which lasts approximately one hour. The third visit involves drawing blood for laboratory testing and blood banking for future lab studies, lasting roughly 4 hours. The glucose tolerance test is administered. The fourth and final visit is an assessment of the participant's metabolism and exercise testing. This visit lasts approximately two hours.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 years or older
* Healthy male or female
* Normal control volunteers and early Alzheimer's disease patients
* Clinical Dementia Rating of 0, 0.5, or 1.0
* On stable doses of medications

Exclusion Criteria:

* Unstable angina
* Schizophrenia
* Clinical signs of depression; major depression; mental health disorder; nervous system disorder
* Significant visual/auditory impairment
* Significant system illness; cancer
* Pacemaker/metal
* Thyroid problems
* Kidney dialysis
* Organ transplant
* Alcoholism
* Heart surgery
* Insulin

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: KU memory clinic patients, volunteers from the community, and the states of Kansas and Missouri
Sampling Method: Non-Probability Sample
Enrollment: 172 (Actual)
Dates: Start 2004-11 (Actual); Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Burns, MD, Principal Investigator — University of Kansas Medical Center, Landon Center on Aging
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States